CLINICAL TRIAL: NCT02458209
Title: A Phase 1, Open-label, Randomized, Single Dose, Parallel Group Comparability Study To Assess The Subcutaneous Pharmacokinetics And Pharmacodynamics Of Bococizumab In Healthy Adult Subjects For Comparisons Of Drug Substance Manufactured At Two Different Locations And Administration Via Prefilled Syringe Vs. Prefilled Pen
Brief Title: Single Dose Manufacturing Site (Pfizer vs. BIP) And Device (Prefilled Syringe vs. Prefilled Pen) Comparability Study For Bococizumab In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B1481026
Record Dates: First submitted 2015-05-01; First posted 2015-06-01 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: PK, bococizumab, comparability, LDL-C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Active Comparator): 150 mg SC dose administered in a prefilled syringe using drug substance manufactured at Pfizer Andover
  Interventions: Biological: bococizumab PFS:Pfizer
- Treatment B (Experimental): • Treatment B: 150 mg SC dose administered in a prefilled syringe using drug substance manufactured at Boehringer Ingelheim Pharma
  Interventions: Biological: bococizumab PFS: BIP
- Treatment C (Experimental): 150 mg SC dose administered in a prefilled pen using drug substance manufactured at Pfizer Andover.
  Interventions: Biological: bococizumab PFP

INTERVENTIONS:
Biological: bococizumab PFS:Pfizer — 150 mg bococizumab administered SC in a prefilled syringe using drug substance manufactured at Pfizer Andover
  Arms: Treatment A
Biological: bococizumab PFS: BIP — 150 mg bococizumab administered SC in a prefilled syringe using drug substance manufactured at Boehringer Ingelheim Pharma.
  Arms: Treatment B
Biological: bococizumab PFP — 150 mg bococizumab administered SC in a prefilled pen using drug substance manufactured at Pfizer Andover
  Arms: Treatment C

SUMMARY:
This is an open label, single dose, randomized, parallel group study in healthy adult subjects to assess the comparability of bococizumab administered in a prefilled syringe vs. prefilled pen and comparability between drug substance manufactured at Pfizer Andover vs. Boehringer Ingelheim Pharma.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and/or female subjects between the ages of 18 and 65 years
2. Body Mass Index (BMI) 33.0 kg/m2 or lower; and a total body weight 60 to 90 kg (132 198 lbs) inclusive
3. Fasting LDL-C must be 80 to 200 mg/dL at two qualifying visits: initial screening (Days -28 to -14) and Day -7.
4. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
5. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant disease or other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results
2. Any condition possibly affecting drug absorption.
3. Pregnant/breast feeding female subjects; male subjects with partners currently pregnant; male & female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception
4. History of allergic or anaphylactic reaction to any therapeutic or diagnostic mAb or molecules made of components of mAb
5. History of regular alcohol consumption : >7 drinks/wk (F) or 14 drinks/wk (M)
6. History of sensitivity to heparin or heparin-induced thrombocytopenia.
7. Positive urine drug screen.
8. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
9. Screening seated BP of 140/90 mm Hg or higher
10. Screening 12-lead ECG demonstrating QTc >450 or a QRS interval >120 msec
11. Subjects with prior exposure to bococizumab (also known as PF-04950615 or RN316) or other investigational PCSK9 inhibitors.
12. Treatment with marketed or investigational mAbs within 6 months or 5 half-lives of Day 1
13. Treatment with an investigational drug within 30 days or 5 half-lives of Day 1, and/or anticipated to take part in a clinical study during the duration of this study.
14. Use of prescription or nonprescription drugs within 7 days or 5 half-lives of Day 1;
15. Abnormal labs:

    AST/SGOT or ALT/SGPT greater than or equal to 1.2 × ULN; total bilirubin greater than or equal to 1.5 × ULN; CK >1.5 × ULN or absolute value >600 U/L.
16. Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
17. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 - Day 85
  maximal plasma concentration
AUCinf | Day 1 - Day 85
  area under the concentration time curve from time 0 extrapolated to infinite time (AUCinf)
Cmax for bococizumab using DS from Pfizer as comapred to DS from BIP | Day 1 - Day 85
  Cmax of bococizumab using drug substance (DS) manufactured by Pfizer vs. DS manufactured by BIP
AUCinf for bococizumab using DS from Pfizer as comapred to DS from BIP | Day 1 - Day 85
  Cmax of bococizumab using drug substance (DS) manufactured by Pfizer vs. DS manufactured by BIP
Cmax for bococizumab using PFS as comapred to PFP | Day 1 - Day 85
  Cmax of bococizumab administered via prefilled syringe vs. a prefilled pen
AUCinf for bococizumab using PFS as comapred to PFP | Day 1 - Day 85
  AUcinf of bococizumab administered via prefilled syringe vs. a prefilled pen

SECONDARY OUTCOMES:
MaxELDL-C | Day 1 - Day 85
  Maximum lowering in LDL C
AUEClast | Day 1 - Day 85
  Area under the LDL C concentration time profile from time zero to the time of the last quantifiable concentration (Clast)
Tmax,LDL-C | Day 1 - Day 85
  Time for MaxELDL- C
Tmax | Day 1 - Day 85
  Time to Cmax
CL/F | Day 1 - Day 85
  apparent clearance
Vz/F | Day 1 - Day 85
  Apparent volume of distribution
T1/2 | Day 1 - Day 85
  terminal half-life
AUClast | Day 1 - Day 85
  Area under the concentration time curve from time 0 to the time of last quantifiable concentration
Incidence of ADAs and neutralizing antibodies | Day 1 - 85
  Incidence of anti-drug antibodies and neutralizing antibodies (if applicable).
Titer for ADAs and neutralizing antibodies | Day 1 - 85
  Titer for anti-drug antibodies and neutralizing antibodies (if applicable).
Incidence, severity and causal relationship of treatment emergent AEs | Day 1 - 85
  Incidence, severity and causal relationship of treatment emergent AEs (TEAEs)
Incidence and severity of ISRs | Day 1 - 85
  Incidence, and severity of injection site reactions
Incidence of abnormal and clinically relevant safety laboratory parameters | Day 1 - 85
  Incidence of abnormal and clinically relevant safety laboratory tests including clinical chemistry, hematology, and vital signs.
MaxELDL-C using DS from Pfizer as compared to BIP, if applicable | Day 1 - Day 85
  Maximum lowering in LDL-C using DS manufactured by Pfizer vs. BIP, if applicable
AUEClast using DS from Pfizer as compared to BIP, if applicable | Day 1 - Day 85
  Area under the LDL-C curve using DS manufactured by Pfizer vs. BIP, if applicable
MaxELDL-C using PFS as compared to PFP, if applicable | Day 1 - Day 85
  Maximum lowering in LDL-C using prefilled syringe vs. prefilled pen , if applicable
AUEClast using PFS as compared to PFP, if applicable | Day 1 - Day 85
  Area under the LDL-C curve using prefilled syringe vs. prefilled pen , if applicable

OTHER OUTCOMES:
PCSK9 | Day 1 - Day 85
  on trial ng/mL PCSK9 concentration, ng/mL change from baseline and percent change from baseline in PCSK9 following bococizumab administration
total cholesterole | Day 1 - Day 85
  on trial mg/mL total cholesterol concentration, change from baseline and percent change from baseline in total cholesterol following bococizumab administration
HDL-C | Day 1 - Day 85
  on trial mg/mL HDL-C concentration, change from baseline and percent change from baseline in HDL-C following bococizumab administration
Non HDL-C | Day 1 - Day 85
  on trial mg/mL non HDL-C concentration, change from baseline and percent change from baseline in non HDL-C following bococizumab administration
triglyceride | Day 1 - Day 85
  on trial mg/mL triglyceride concentration, change from baseline and percent change from baseline in triglyceride following bococizumab administration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Broward Research Group, Hollywood, Florida
  - Miami Research Associates, LLC, South Miami, Florida
  - MRA Clinical Research, LLC, South Miami, Florida
  - Prism Research, LLC, Saint Paul, Minnesota
  - High Point Clinical Trials Center, LLC, High Point, North Carolina

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] Wang EQ, Plotka A, Salageanu J, Baltrukonis D, Mridha K, Frederich R, Sullivan BE. Comparative Pharmacokinetics and Pharmacodynamics of Bococizumab Following a Single Subcutaneous Injection Using Drug Substance Manufactured at Two Sites or Administration via Two Different Devices. Clin Pharmacol Drug Dev. 2019 Jan;8(1):40-48. doi: 10.1002/cpdd.454. Epub 2018 Apr 24. PMID 29688615
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481026&StudyName=A%20Phase%201%2C%20Open-label%2C%20Randomized%2C%20Single%20Dose%2C%20Parallel%20Group%20Comparability%20Study%20To%20Assess%20The%20Subcutaneous%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Bococizumab%20In%20Healthy%20Adult%20Subjects%20For%20Comparisons%20Of%20Drug%20Substance%20Manufactured%20At%20Two%20Different%20Locations%20And%20Administration%20Via%20Prefilled%20Syringe%20Vs.%20Prefilled%20Pen